CLINICAL TRIAL: NCT05444478
Title: Microwave Ablation Simultaneously Combined With Lenavatinib for Recurrent Hepatocellular Carcinoma: a Prospective Randomized Controlled Study
Brief Title: Microwave Ablation Simultaneously Combined With Lenavatinib for Recurrent Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect 2
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma; Microwave Ablation; Liver Cancer; Lenvatinib; Recurrent Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Recurrence | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave ablation (Experimental): Patients only accepted microwave ablation
  Interventions: Procedure: Microwave ablation
- Microwave ablation plus lenvatinib (Experimental): Patients accepted microwave ablation plus lenvatinib
  Interventions: Procedure: Microwave ablation; Drug: Lenvatinib

INTERVENTIONS:
Procedure: Microwave ablation — only microwave ablation for tumor
Drug: Lenvatinib — lenvatinib (80 mg for body no more than 60kg，120 mg for body weight >60 kg)
  Arms: Microwave ablation plus lenvatinib

SUMMARY:
This study intends to evaluate the efficacy and safety of microwave ablation combined lenvatinib simultaneously for recurrent HCC

DETAILED DESCRIPTION:
Microwave ablation (MWA) is available as the major curative treatments for early-stage recurrent HCC. Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma. No study has evaluated MWA simultaneously combined Lenvatinib for recurrent HCC. There needs further investigation to explore the efficacy and safety of the combination treatment. Thus, the investigators carried out this randomized, multicenter, prospective trial study to find out it.

ELIGIBILITY:
Inclusion Criteria:

1. Primary HCC (BCLC 0-B), and the pathological results is hepatocellular carcinoma；
2. recurrent HCC without any tumor related therapy；
3. Tumor number ≤3；
4. Tumor size ≤5cm;
5. Good performance, KPS≥90；
6. Age：18-75
7. Child-Pugh A or B（score of the B level is no more than 7）
8. Baseline laboratory examinations meet the Criteria： Leukocyte ≥3.0×109/L； Blood platelet ≥75×109/L； Hemoglobin ≥100g/L； ALT、AST ≤ 3 x limit of normal（ULN）； Serum creatinine ≤ 1.5 x ULN； Prothrombin time < ULN+4 s；INR < 1.5, Albumin ≥30g/L ； Total bilirubin ≤34mmol/L；

Exclusion Criteria:

1. disagreeing to receive follow-up observation and participate the clinical study;
2. Accompanying with a history of other malignancies;
3. Accompanying with macrovascular invasion such as portal vain tumor thrombus, hepatic vein tumor thrombus;
4. with extrahepatic metastasis or lymph metastasis;
5. receiving system therapy such as targeted therapy or immunotherapy;
6. receiving local therapy such as ablation or TACE;
7. Any of the following occurred within 12 months of the study: myocardial infarction, severe / unstable angina, coronary artery bypass grafting, congestive heart failure, cerebrovascular accident (including transient ischemic attack), pulmonary embolism; ongoing arrhythmia by NCI-CTCA standard ≥ 2, prolonged QTc interval (450 ms for males, and> 470 ms for females;
8. other serious acute, chronic physiological or mental disorders or abnormal laboratory examination may increase the risk of participation in study treatment or may interfere with the interpretation of study findings or whom the investigator considers not fit;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Tumor-free survival rate at 36 months | 36 months
  Progression was defined as progressive disease after microwave ablation by independent radiologic review according to mRECIST or death from any cause
Over-all survival (OS) rate at 36 months | 36 months
  OS is the length of time from the date of microwave ablation until death from any cause.

SECONDARY OUTCOMES:
Adverse events | 24 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.
Complication rate | 36 months
  Complication was defined as the a disease or sythrome caused by the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xianhai Mao, Professor, Study Director — Hunan Provincial People's Hospital
Locations (1):
- Hunan Provincial People's Hospital, Changsha, Hunan, China